CLINICAL TRIAL: NCT02870036
Title: Study to Evaluate the Safety, Tolerability, Preliminary Efficacy and Pharmacokinetics of Simmitecan Monotherapy and Combination in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GV-LP-102
Record Dates: First submitted 2016-08-03; First posted 2016-08-17 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Advanced Solid Tumor; Advanced/Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — simmitecan; Fluorouracil; Leucovorin; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Pharmacokinetic data investigation of Simmitecan (Experimental): To further determine the pharmacokinetic (PK) characteristics of Simmitecan monotherapy in patients with advanced solid tumors
  Interventions: Drug: Simmitecan
- Dose escalation study of Simmitecan combined therapy (Experimental): To determine the maximum tolerated dose (MTD) of Simmitecan combined with 5-fluorouracil/Leucovorin Calcium in patients with advanced solid tumor
  Interventions: Drug: Simmitecan; Drug: 5-fluorouracil and Leucovorin Calcium
- Dose extension study of Simmitecan monotherapy (Experimental): To preliminarily evaluate the anti-tumor activity of Simmitecan monotherapy in patients with advanced solid tumors, and to determine the recommended phase II dose (RP2D)
  Interventions: Drug: Simmitecan
- Dose extension study of Simmitecan combined Thalidomide (Experimental): To preliminarily evaluate the anti-tumor activity of Simmitecan combined with 5-fluorouracil/Leucovorin Calcium in patients with advanced/metastatic colorectal cancer (CRC), and to determine RP2D
  Interventions: Drug: Simmitecan; Drug: Thalidomide
- Dose escalation&extension Simmitecan combined Thalidomide (Experimental): To preliminarily evaluate the anti-tumor activity of Simmitecan combined with thalidomide in patients with gastrointestinal tumors, and to determine RP2D and MTD
  Interventions: Drug: Simmitecan; Drug: Thalidomide
- Dose extension study of Simmitecan combined therapy (Experimental): To preliminarily evaluate the anti-tumor activity of Simmitecan combined with thalidomide in patients with specific tumors
  Interventions: Drug: Simmitecan; Drug: 5-fluorouracil and Leucovorin Calcium

INTERVENTIONS:
Drug: Simmitecan
Drug: 5-fluorouracil and Leucovorin Calcium
  Arms: Dose escalation study of Simmitecan combined therapy; Dose extension study of Simmitecan combined therapy
Drug: Thalidomide
  Arms: Dose escalation&extension Simmitecan combined Thalidomide; Dose extension study of Simmitecan combined Thalidomide

SUMMARY:
This study evaluates the safety, tolerability, preliminary efficacy and pharmacokinetics of Simmitecan in patients with advanced solid tumors and Simmitecan, 5-fluorouracil and Leucovorin Calcium,thalidomide in patients with advanced solid tumor or advanced/metastatic colorectal cancer.

ELIGIBILITY:
Inclusion criteria

1. Patients who have fully understood the study, and are willing to sign the informed consent (ICF);
2. Patients with advanced solid tumor confirmed by histopathology and/or cytology were enrolled in Parts 1 and 2 of the study; Four groups of patients with advanced solid tumor confirmed by histopathology and/or cytology were enrolled in Part 3 of the study: Group 1 consisted of patients with rectal carcinoma, Group 2 consisted of patients with gastric carcinoma and esophageal carcinoma, Group 3 consisted of patients with biliary duct carcinoma and pancreatic carcinoma, and Group 4 consisted of patients with gastro-entero-pancreatic neuroendocrine carcinoma. Patients with advanced or metastatic CRC confirmed by histopathology and/or cytology were enrolled in Part 4 of the study; In Part 5 of the study, patients with advanced gastrointestinal tumor (including biliary tumor [gallbladder carcinoma, intra- or extra-hepatic biliary carcinoma], pancreatic carcinoma, hepatocellular carcinoma, esophageal carcinoma, gastric carcinoma, colorectal carcinoma, gastrointestinal stromal carcinoma, and gastro-entero-pancreatic neuroendocrine carcinoma) confirmed by histopathology were enrolled; In Part 6 of the study, patients with advanced gastrointestinal tumor (tentatively determined as biliary tumor, hepatocellular carcinoma, pancreatic carcinoma, and colorectal carcinoma); At least 5 unstained slices of tumor tissues must be obtained at baseline from patients participating in Parts 5 and 6 of the study: Primary lesion samples at the initial diagnosis or archived recently were acceptable. They were used to detect protein expression level of SOD1 and other related molecules to and tumor immunity related indicators.

   Note: patients being enrolled in part 2 of the study should be those with advanced solid tumor who are suitable for therapeutic regimen of Simmitecan combined with 5 FU/LV as judged by the investigator;
3. Patients who had failed standard treatments for advanced cancer, or are intolerant to the current standard treatments, or no suitable standard treatments available for advanced cancer;
4. Patients who have at least one measurable lesion (according to RECIST, version 1.1); note: the lesions previously treated with radiotherapy cannot be regarded as the target lesion, unless the lesion showed clear progression after radiotherapy;
5. Patients with Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
6. Age≥ 18 years and ≤ 70 years, male or female is allowed;
7. Patients with life expectancy of 12 weeks or more;
8. Patients with appropriate organ function as documented by:

   1. absolute neutrophil count ≥ 1.5 × 109/L;
   2. hemoglobin ≥ 9 g/dL (without RBC transfusion within 14 days);
   3. platelet count ≥ 100 × 109/L.
   4. serum total bilirubin ≤1.5 times of upper limit of normal (ULN) (for the patients with Gilbert syndrome, total bilirubin is allowed to be ≤ 3 × ULN and direct bilirubin is allowed to be 1.5 × ULN);
   5. aspertate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN, or AST and ALT ≤ 5 × ULN for patients with liver metastasis;
   6. creatinine clearance ≥ 50 mL/min (calculated by MDRD equation, see appendix 7);
   7. international normalized ratio (INR) ≤1.5 × ULN, or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (INR only for patients who were not given anticoagulant therapy).
9. Patients with negative hepatitis b surface antigen; for patients with positive hepatitis b surface antigen, quantitative result of hepatitis b virus (HBV) DNA should be lower than 1000 cps/mL;
10. Toxicity events caused by previous treatments, surgery or radiotherapy have recovered to CTCAE grade 0 or 1 (except for alopecia);
11. Female patients are eligible for the study if the following conditions are met:

    1. Patients have no fertility (i.e., physiological infertility), including postmenopausal period (complete menolipsis for more than 1 year) or documented irreversible sterilization operation including hysterectomy, bilateral ovariectomy, or bilateral salpingectomy (instead of tubal ligation);
    2. For patients of childbearing potential, the results of serum pregnancy test screening should be negative (within 7 days before the first dose of investigational drug), and breastfeeding is not allowed before the start of the study and throughout the study. Moreover, the patients should agree to take effective contraception measures during the study and within 90 days after the last dose, and should always conduct strict birth control in accordance with the label of drug/appliance and the investigator's instructions. Effective contraception measure is defined as:

       * The sexual partner with removed deferens is the only sexual partner of female patient;
       * Use of any intrauterine device with documented failure rate less than 1% per year;
       * Double contraception, such as spermicide plus male condom, female condom, diaphragm, cervical cap or intrauterine contraceptive device.
12. Male patients should have undergone vasectomy, or agree to take effective contraception measures during the study and within 90 days after the last dose;
13. Patients are able to follow the study procedures, restrictions and requirements at the investigator's discretion.

Exclusion criteria

1. Patients are still within 5 half-life of previous anticancer chemotherapy, biological agents or other investigational drugs (if 5 half-life exceeds 28 days, calculated as 28 days) at the time of screening;
2. Patients received systemic radiotherapy (including whole brain radiotherapy) within 28 days before enrollment, or received small area radiotherapy (stereotactic radiotherapy of central nervous system (CNS)) within 7 days before enrollment, or have not yet recovered from the previous radiotherapy;
3. Patients have not yet recovered from the toxic effects (except alopecia) caused by previous anti-tumor treatments (> CTCAE grade 1);
4. Patients underwent major surgery or have not yet been fully recovered from pervious surgery (major surgery is defined as grade 3 or 4 surgery specified in "Management Measures for Clinical Application of Medical Technology" implemented on May 1st, 2009).
5. Patients had CNS metastasis or cancer-related epilepsy requiring clinical intervention; however, patients with CNS metastasis who received treatments, or the asymptomatic patient can be enrolled;
6. Patients with a history of allergy to 5-FU or LV;
7. Patients with active HBV or HCV infection;
8. Patients diagnosed as human immunodeficiency virus (HIV) infection, or are not willing to have HIV test;
9. Patients with clinically significant active infection;
10. Patients with previous or concurrent other malignant tumors (except effectively controlled non-melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ, and other effectively controlled tumors in the past 5 years even without treatments);
11. Patients with impaired cardiac function or clinically significant heart diseases, including grade 2 or higher congestive heart failure per New York Heart Association (NYHA) classification, arrhythmia, conduction abnormalities requiring treatment, cardiomyopathy, or uncontrolled hypertension;
12. Patients with serious kidney damage requiring kidney dialysis;
13. Patients with serious liver damage, grade B or C end-stage liver diseases per Child-Pugh classification (see appendix 8);
14. Any other diseases or conditions with clinical significance that may affect the protocol compliance or patient's signature of ICF at the investigator's discretion (such as uncontrolled diabetes, etc.);
15. Patients with disease of digestive tract such as duodenal ulcer, ulcerative colitis, intestinal obstruction or other conditions that may cause alimentary tract hemorrhage or perforation as judged by the investigator, or have past medical history of gastric-intestinal perforation or intestinal fistula;;
16. Patient's physical condition cause the risk of investigational drug use, or render the toxicity or AE difficult to explain at the investigator's discretion.
17. Patients who received Irinotecan therapy within 3 months prior to enrollment.
18. Patients with arteriovenous thromboembolic events within the past 6 months, including myocardial infarction, cerebral stroke, deep vein thrombosis, or pulmonary embolism, etc.
19. Patients who were sensitive to Thalidomide (in Parts 5 and 6).
20. Peripheral neuropathy CTCAE ≥ Grade 2 (in Parts 5 and 6).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cmax (maximum plasma concentration) | before administration (within 5 minutes before administration), 45 and 90 minutes after the start of the infusion of Simmitecan and at 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48 and 72 hours after the completion of infusion of Simmitecan
Tmax (time to maximum plasma concentration) | before administration (within 5 minutes before administration), 45 and 90 minutes after the start of the infusion of Simmitecan and at 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48 and 72 hours after the completion of infusion of Simmitecan
AUC (area under the plasma concentration-time curve) | before administration (within 5 minutes before administration), 45 and 90 minutes after the start of the infusion of Simmitecan and at 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48 and 72 hours after the completion of infusion of Simmitecan
T½ | before administration (within 5 minutes before administration), 45 and 90 minutes after the start of the infusion of Simmitecan and at 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48 and 72 hours after the completion of infusion of Simmitecan
CL (systemic clearance) | before administration (within 5 minutes before administration), 45 and 90 minutes after the start of the infusion of Simmitecan and at 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48 and 72 hours after the completion of infusion of Simmitecan
Vz (apparent volume of distribution) | before administration (within 5 minutes before administration), 45 and 90 minutes after the start of the infusion of Simmitecan and at 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48 and 72 hours after the completion of infusion of Simmitecan
Adverse events (AE) | AEs will be classified by type, incidence, severity (graded per NCI-CTCAE [version 4.03]), time to onset, seriousness and relationship

SECONDARY OUTCOMES:
Objective response rate (ORR) | Imaging examination will be performed for tumor assessment every 6 weeks (±7 days) from the first dose of Simmitecan until PD, intolerable toxicity, withdrawal of consent or death.
  Tumor will be evaluated according to RECIST-1.1. CT or MRI can be used for tumor imaging at the investigator's discretion.
progression free survival (PFS) | Imaging examination will be performed for tumor assessment every 6 weeks (±7 days) from the first dose of Simmitecan until PD, intolerable toxicity, withdrawal of consent or death.
  Tumor will be evaluated according to RECIST-1.1. CT or MRI can be used for tumor imaging at the investigator's discretion.
CBR (clinical benefit rate) | Imaging examination will be performed for tumor assessment every 6 weeks (±7 days) from the first dose of Simmitecan until PD, intolerable toxicity, withdrawal of consent or death.
  Tumor will be evaluated according to RECIST-1.1. CT or MRI can be used for tumor imaging at the investigator's discretion.
DCR (disease control rate) | Imaging examination will be performed for tumor assessment every 6 weeks (±7 days) from the first dose of Simmitecan until PD, intolerable toxicity, withdrawal of consent or death.
  Tumor will be evaluated according to RECIST-1.1. CT or MRI can be used for tumor imaging at the investigator's discretion.
OS (overall survival) | Imaging examination will be performed for tumor assessment every 6 weeks (±7 days) from the first dose of Simmitecan until PD, intolerable toxicity, withdrawal of consent or death.
  Tumor will be evaluated according to RECIST-1.1. CT or MRI can be used for tumor imaging at the investigator's discretion.
accumulative excretion rate | Accumulative excretion rate within 0-72 h after the first administration of Simmitecan.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Cancer Hospital, Beijin, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tongji Hospital of Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The first hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guimbaud R, Louvet C, Ries P, Ychou M, Maillard E, Andre T, Gornet JM, Aparicio T, Nguyen S, Azzedine A, Etienne PL, Boucher E, Rebischung C, Hammel P, Rougier P, Bedenne L, Bouche O. Prospective, randomized, multicenter, phase III study of fluorouracil, leucovorin, and irinotecan versus epirubicin, cisplatin, and capecitabine in advanced gastric adenocarcinoma: a French intergroup (Federation Francophone de Cancerologie Digestive, Federation Nationale des Centres de Lutte Contre le Cancer, and Groupe Cooperateur Multidisciplinaire en Oncologie) study. J Clin Oncol. 2014 Nov 1;32(31):3520-6. doi: 10.1200/JCO.2013.54.1011. Epub 2014 Oct 6. PMID 25287828
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342